CLINICAL TRIAL: NCT02244294
Title: A Two Phase, Double-blinded, Randomized, Parallel Group Design, Multicenter Study of FLOMAX® Capsules, 0.4 mg Versus Placebo, in Male Patients With Acute Urinary Retention Related to Benign Prostatic Hyperplasia
Brief Title: FLOMAX® Versus Placebo, in Male Patients With Acute Urinary Retention Related to Benign Prostatic Hyperplasia (BPH)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 527.26
Record Dates: First submitted 2014-09-18; First posted 2014-09-19 (Estimated); Last update posted 2014-09-19 (Estimated); Status verified 2014-09

CONDITIONS: Prostate Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Tamsulosin

ARMS (2):
- FLOMAX® (Experimental)
  Interventions: Drug: FLOMAX® capsules
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo capsules

INTERVENTIONS:
Drug: FLOMAX® capsules
  Other Names: Tamsulosin hydrochloride
  Arms: FLOMAX®
Drug: Placebo capsules
  Arms: Placebo

SUMMARY:
To establish whether the administration of FLOMAX® improves the outcome of a trial without catheter (TWOC) after an episode of acute urinary retention and to determine whether spontaneous voiding is maintained over the course of six months of active treatment

ELIGIBILITY:
Inclusion Criteria:

Phase I

* Adult men, 45 years of age or older, diagnosed with acute urinary retention due to BPH
* Patients who have never taken alpha-blockers or discontinued taking alpha-blockers 72 hours or more prior to entrance into this study
* Patients that have been treated with an indwelling urethral catheter as treatment for acute urinary retention (AUR) due to BPH
* Patients must be judged by the investigator to be reliable and willing to comply with all tests and examinations stipulated in the protocol
* All patients must be willing to give meaningful, written, informed consent prior to participation in the trial, in accordance with regulatory requirements. Patients must also have sufficient understanding to communicate effectively with the investigator

Phase II - Patients who voided spontaneously, at least 100 mL and a post-void residual volume of ≤ 300 mL, at Visit 2

Exclusion Criteria:

Phase I

* Patients diagnosed with a symptomatic/active urinary tract infection (UTI) or an abnormal urine culture at baseline or 2 or more UTIs within the last six months. An abnormal urine culture was defined as:

  * A bacterial colony count of greater than or equal to 100,000 CFU/mL or
  * A bacterial colony count of greater than or equal to 100 CFU/mL of a known urinary pathogen in a symptomatic patient
* Patients that have a distended bladder volume greater than 1.5 liters (1500 ml) of retention as measured by initial catheter urine volume
* Patients with history of sexually transmitted disease within last two years
* Patients with active genital herpes disease whose urinary function was impacted due to the disease
* Patients who have a history of mechanical outlet obstruction excluding BPH (i.e., bladder neck contracture or stricture, bladder tumor, or bladder calculi)
* Patients with urethral stricture disease
* Patients with a history of bladder, prostate, or urethral surgery in the last three months
* Patients presenting with AUR who were not been seen within 5 days of urethral catheter placement
* Patients presenting with any of the following: active urinary stone disease, previous pelvic radiotherapy, perirectal inflammatory disorders or inflammatory bowel disease
* Participation in another drug study within 30 days of Visit 1
* Clinically relevant conditions which may interfere with the patient's ability to participate in the study including, but not limited to, the following: neurologic, gastrointestinal, cardiovascular, hepatic, renal, psychiatric, hematologic or respiratory disease and clinically relevant laboratory abnormalities not mentioned above (e.g., hematuria) based upon the clinical judgment of the investigator
* Patients receiving cimetidine, ranitidine or warfarin within two weeks of study start date and who would potentially use such medications during the course of the trial
* Patients currently treated with finasteride (PROSCAR®) and who would not discontinue its use upon entrance into the study
* Patients with known hypersensitivity to FLOMAX® (tamsulosin hydrochloride) or other alpha-blockers
* Patients with a history of myocardial infarction within six months of baseline
* Patients with uncontrolled hypertension (systolic > 160 mmHg, diastolic > 100 mmHg) and patients with severe hypotension (systolic < 90 mmHg)
* Patients who have been using the following drugs, 72 hours prior to study start date, or who are unable to discontinue these drugs over the course of the study:

  * Alpha-adrenergic medication
  * Drugs with systemic anticholinergic activity including antihistamines. The following antihistamines are allowed: ALLEGRA®, CLARITIN® or ZYRTEX®
  * Antispasmodics or muscle relaxants
  * Parasympathomimetics, cholinomimetics or similar drug
* Patients that have poorly controlled diabetes mellitus who suffer from peripheral neuropathy or diabetic cystopathy
* Patients who suffer from neurological diseases affecting the bladder (i.e., multiple sclerosis, Parkinson's disease, stroke, and any bladder trauma that may be an exclusion criterion in the opinion of the investigator
* Patients with a neurological impairment or psychiatric disorder that prevents their comprehension of the informed consent and/or the ability to comply with the protocol
* Patients with a urine volume at the initial catheterization less than 300 mL
* Patients with a diagnosis of active cancer, except basal cell carcinoma, within 5 years or less
* Patients who had a transurethral resection of the prostate (TURP) within 5 years or less of study enrollment and irreversible urethral damage due to the procedure

Phase II

- Patients with clinically, significant abnormal lab results including any baseline laboratory serum test with the following values:

* Hemoglobin < 11.0 g/dL
* Leukocytes < 3,000 per mm3
* Liver enzymes [aspartate aminotransferase (SGOT), alanine transaminase (SGPT) and alkaline phosphatase]: more than two times the upper limit of normal at baseline
* Serum creatinine more than two times the upper limit of normal at Visit 1
* Patients with clot retention, persistent gross hematuria (Visit 3 only), prostatitis, a symptomatic/active urinary tract infection (UTI) or an abnormal baseline urine culture
* An abnormal urine culture was defined as:
* A bacterial colony count of greater than or equal to 100,000 colony forming units (CFU)/mL or
* A bacterial colony count of greater than or equal to 100 CFU/mL of a kown urinary pathogen in a symptomatic patient

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2001-03; Primary Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Successful spontaneous voiding after urethral catheter removal | Up to 96 hours after start of treatment
  For Phase I of the trial
Maintenance of successful spontaneous voiding | Up to 6 months after start of treatment
  For Phase II of the trial

SECONDARY OUTCOMES:
Change in voided urine volume | Up to 6 months after start of treatment
Determination of post-void residual urine volume | Up to 6 months after start of treatment
  by ultrasound or bladder scan
Time to recurrence of AUR | Up to 6 months after start of treatment
  For phase II of the trial
Clinically significant changes from baseline in vital signs | Pre-dose, up to 6 months after start of treatment
Number of patients with adverse events | Up to 6 months